CLINICAL TRIAL: NCT03233022
Title: A Randomized Trial Examining the Impact of Five 8-week Online Well-being Programs on Mood and Well-being
Brief Title: An Online Trial of Five Well-being Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Happify Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2017-08

CONDITIONS: Well-being

STUDY DESIGN:
Intervention Model Description: Users are randomly assigned between arms after completing baseline assessment and stay in that arm for the duration of the study.
Oversight: Data Monitoring Committee: No

ARMS (5):
- Unchanged Happify (Active Comparator): Participants use Happify as it is currently available to consumers on the main site, including all engagement elements. Users may access a wide variety of 4-week programs and use them in any way they desire for the entire study period.
  Interventions: Behavioral: Happify
- Negatively-focused tracks (Active Comparator): Participants use two pre-selected Happify tracks that focus on remediating negatives (e.g. "conquering negative thoughts" and "managing stress"). Several engagement elements are missing, including social forums, regular informational emails, and the ability to play games. Participants gain access to 8 weeks worth of content, but may repeat the content as often as they like in the follow-up period.
  Interventions: Behavioral: Happify
- Positively-focused tracks (Active Comparator): Participants use two pre-selected Happify tracks that focus on improving positives (e.g. building well-being, using one's strengths). Several engagement elements are missing, including social forums, regular informational emails, and the ability to play games. Participants gain access to 8 weeks worth of content, but may repeat the content as often as they like in the follow-up period.
  Interventions: Behavioral: Happify
- Placebo condition (Placebo Comparator): Participants complete a Happify program that is designed to engage with specific activities, but that does not aim to promote positive emotion or reduce negative emotion. Participants gain access to 8 weeks worth of content, but may repeat the content as often as they like in the follow-up period.
  Interventions: Behavioral: Happify
- Distraction condition (Sham Comparator): Participants complete a series of quizzes and polls on Happify designed to engage them in thinking about well-being topics, but without giving any specific instructions for how to promote well-being. Participants gain access to 8 weeks worth of content, but may repeat the content as often as they like in the follow-up period.
  Interventions: Behavioral: Happify

INTERVENTIONS:
Behavioral: Happify — An online platform for conveying techniques from positive psychology, cognitive-behavioral therapy, and mindfulness-based stress reduction.

SUMMARY:
Participants complete an 8-week program and complete assessment measures to track their outcomes over time.

DETAILED DESCRIPTION:
Participants will be randomly assigned between five different well-being programs, each 8-weeks long and taking place on a simplified research version of the Happify platform. They will be asked to complete questionnaires before and after the 8-week program, as well as 1-month, 3-month, and 6-month follow-up questionnaires after the program is complete, at which point study participation will end.

ELIGIBILITY:
Inclusion Criteria:

* No prior experience on the Happify platform (new user registration)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14000 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms (Patient Health Questionnaire 9-item; PHQ-9) | Change from baseline to 8-week post, 1-month, 3-month, and 6-month follow-up
  9-item measure of depressive symptoms
Anxiety Symptoms (Generalized Anxiety Disorder 7-item; GAD-7) | Change from baseline to 8-week post, 1-month, 3-month, and 6-month follow-up
  7-item measure of anxiety symptoms

SECONDARY OUTCOMES:
Resilience composite | Change from baseline to 8-week post, 1-month, 3-month, and 6-month follow-up
  Composite score made of perceived stress, positive emotionality, and optimism

CONTACTS AND LOCATIONS:
Locations (1):
- Happify (an online platform -- study is entirely online), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carpenter J, Crutchley P, Zilca RD, Schwartz HA, Smith LK, Cobb AM, Parks AC. Seeing the "Big" Picture: Big Data Methods for Exploring Relationships Between Usage, Language, and Outcome in Internet Intervention Data. J Med Internet Res. 2016 Aug 31;18(8):e241. doi: 10.2196/jmir.5725. PMID 27580524
- See also: Site where study is taking place. — http://www.happify.com